CLINICAL TRIAL: NCT07288866
Title: Effect of the Use of Oocyte-specific or Universal Vitrification and Warming Media on Pregnancy Rates in the Context of Oocyte Donation
Brief Title: Effect of Vitrification and Warming Media on Pregnancy Rates in the Context of Oocyte Donation
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2025_BRUGNON
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2024-04

CONDITIONS: Infertility; Infertility, Female
Keywords: Cryopreservation; Cryobiology; Vitrification; Oocyte donation; Cryoprotective Agents
MeSH Terms: conditions — Infertility; Infertility, Female | interventions — Vitrification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- S/S - Vitrified and warmed with Oocyte-specific medium: 41 oocyte recipient ICSI cycles for which the initial oocyte vitrification procedure was performed with "oocyte- specific" medium RapidVit™ Oocyte (Vitrolife) and the warming procedure was performed with "oocyte-specific" medium RapidWarm™ Oocyte (Vitrolife)
  Interventions: Other: Vitrification and warming media for oocyte vitrification
- S/U - Vitrified with Oocyte-specific medium, Warmed with universal medium: 39 oocyte recipient ICSI cycles for which the initial oocyte vitrification procedure was performed with "oocyte- specific" medium RapidVit™ Oocyte (Vitrolife) and the warming procedure was performed with "universal" medium RapidWarm™ Omni (Vitrolife)
  Interventions: Other: Vitrification and warming media for oocyte vitrification
- U/U - Vitrified and warmed with universal medium: 31 oocyte recipient ICSI cycles for which the initial oocyte vitrification procedure was performed with "universal" medium RapidVit™ Oocyte (Vitrolife) and the warming procedure was performed with "universal" medium RapidWarm™ Omni (Vitrolife)
  Interventions: Other: Vitrification and warming media for oocyte vitrification

INTERVENTIONS:
Other: Vitrification and warming media for oocyte vitrification — Different combinations of the vitrification and warming media were used for oocyte vitrification procedure in the context of oocyte donation

SUMMARY:
Vitrification has become the gold standard for oocyte and embryo cryopreservation. Several commercial kits are available on the market, some are designed for specific developmental stages (e.g. oocytes, zygotes, cleavage-stage embryos or blastocysts) and others are suitable for several stages, therefore termed "universal". Oocytes, cleavage-stage embryos and blastocysts display different levels of resistance to cryopreservation, due to stage-specific properties. While the composition and the exposition protocol of stage specific media are optimized for specific developmental stages, "universal" media display a single composition, therefore exposition protocols should be adapted to each specific developmental stage to ensure optimal survival rates.

The main objective of this study is to determine whether the shift from "oocyte specific" vitrification and warming media to "universal" media has an impact oocyte survival, embryological and clinical outcomes.

DETAILED DESCRIPTION:
A retrospective, monocentric study comparing the clinical and embryological outcomes of 111 oocyte recipient cycles with ICSI from March 2016 to July 2020. Baseline characteristics (donor age and BMI, ovarian stimulation protocol, number of collected oocytes) of the 81 related donations were also analysed.

Two generations of vitrification and warming media were used during this period:

* "Oocyte-specific": RapidVit™ Oocyte and RapidWarm™ Oocyte, Vitrolife
* "Universal": RapidVit™ Omni and RapidWarm™ Omni, Vitrolife Patients were divided in 3 groups according to the combination of the vitrification medium and the warming medium : "specific/specific" (S/S), "specific/universal" (S/U) and "universal/universal" (U/U)..

ELIGIBILITY:
Inclusion Criteria:

* Recipient couples undergoing an oocyte donation ICSI cycle from March 2016 to July 2020 for whom the allocated oocytes were vitrified in our center between July 2015 and January 2020

Exclusion Criteria:

* Recipient couples undergoing an oocyte donation ICSI cycle from March 2016 to July 2020 for whom the allocated oocytes were vitrified prior to July 2015 or after January 2020.

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Oocyte recipient couples undergoing an oocyte donation ICSI
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Impact of vitrification and warming media on clinical pregnancy rate per fresh embryo transfer | UltraSound at 1 month after embryo transfer
  number of clinical pregnancies (one or more gestational sacs visualized in ultrasonography) expressed per 100 embryo transfers

SECONDARY OUTCOMES:
Impact of vitrification and warming media on oocyte survival rate | two hours after warming procedure
  the number of injected oocytes divided by the number of warmed oocytes, expressed as a percentage (%)
Impact of vitrification and warming media on fertilization rate | 16-18 hours
  number of 2PN zygotes divided by the number of injected oocytes, expressed as a percentage (%)
Impact of vitrification and warming media on day-2 embryo percentage | 43-45 hours
  number of cleavage-stage embryos obtained divided by the number of 2PN zygotes, expressed as a percentage (%)
Impact of vitrification and warming media on top-quality embryo percentage | 43-45 hours
  Number of top-quality cleavage-stage embryos obtained divided by the total number of cleavage stage embryos, expressed as a percentage (%).
Impact of vitrification and warming media on blastulation rate | 114-118 hours
  number of blastocysts obtained divided by the number of embryos subjected to extended culture, expressed as a percentage (%)
Impact of vitrification and warming media on good quality blastocyst rate | 114-118 hours
  number of good quality blastocysts (ICM and trophoectoderm grade A or B obtained divided by the total number of blastocysts obtained, expressed as a percentage (%)
Impact of vitrification and warming media on implantation rate | 114-118 hours
  number of gestational sacs with a cardiac activity visualized in ultrasonography divided by the number of embryo transferred, expressed as a percentage (%)
Impact of vitrification and warming media on live birth rate per embryo transfer | 42 weeks
  number live births expressed per 100 embryo transfers
Impact of vitrification and warming media on miscarriage rate per embryo transfer | up to 42 weeks
  number miscarriages expressed per 100 embryo transfers

CONTACTS AND LOCATIONS:
Overall Officials: Florence Brugnon, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France